CLINICAL TRIAL: NCT02020616
Title: Safety, Tolerability, Pharmacokinetics, and Efficacy of LY3053102 With 12 Weeks of Treatment in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of the Safety and Effectiveness of LY3053102 in Participants With Type 2 Diabetes
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of Efficacy
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14515; I6I-MC-LMRB (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-12-13; First posted 2013-12-25 (Estimated); Results first posted 2017-12-20 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- LY3053102 (Experimental): Stage 1: Escalating dose (7 milligrams [mg] up to 200 mg) of LY3053102 administered once a week by subcutaneous (SC) injection for 12 weeks. Stage 2: LY3053102 administered once a week by SC injection for 12 weeks
  Interventions: Drug: LY3053102; Drug: Metformin
- Placebo (Placebo Comparator): Stage 1 and Stage 2: Placebo to match LY3053102 administered by SC injection once a week for 12 weeks
  Interventions: Drug: Placebo; Drug: Metformin
- Exenatide Extended-Release (ER) (Active Comparator): Stage 1 and Stage 2: Exenatide ER 2 mg given by SC injection once a week for 12 weeks
  Interventions: Drug: Exenatide ER; Drug: Metformin
- LY3053102 + Exenatide ER (Experimental): Stage 2: LY3053102 administered by SC injection once a week for 12 weeks and exenatide ER 2 mg administered by SC injection once a week for 12 weeks
  Interventions: Drug: LY3053102; Drug: Exenatide ER; Drug: Metformin

INTERVENTIONS:
Drug: LY3053102 — Administered SC
  Arms: LY3053102; LY3053102 + Exenatide ER
Drug: Exenatide ER — Administered SC
  Arms: Exenatide Extended-Release (ER); LY3053102 + Exenatide ER
Drug: Placebo — Administered SC
  Arms: Placebo
Drug: Metformin — Administered orally (PO)

SUMMARY:
The purpose of this study is to investigate the safety and effectiveness of the study drug known as LY3053102 in participants with Type 2 diabetes mellitus. The study drug will be given in different doses as an injection under the skin. The study is expected to last up to 6 months for each participant. Participants may remain on stable-dose metformin as prescribed by their personal physician.

ELIGIBILITY:
Inclusion Criteria

* Participants with type 2 diabetes mellitus for at least 6 months before entering the trial based on the disease diagnostic criteria (World Health Organization [WHO]) classification managed with diet or exercise alone or with a stable dose of metformin of at least 1000 mg/day for at least 60 days before screening or on metformin and an eligible second oral anti-hyperglycemic medication after a 60-day washout of the second oral anti-hyperglycemic medication
* Women not of childbearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause
* Have a hemoglobin A1c value of ≥7.0% and ≤10.5%, if on diet and exercise or diet, exercise, and metformin (stable dose of at least 1000 mg/day for at least 60 days), or have a hemoglobin A1c value of ≥7.0% and ≤9.5%, and are on an appropriate diet and exercise regimen, a stable dose of metformin and willing to discontinue a second oral anti-hyperglycemic medication
* Have a body mass index ≥23 and ≤45 kilograms per square meter (kg/m^2)

Exclusion Criteria

* Have used insulin for diabetic control for more than 6 consecutive days within 1 year prior to screening
* Have used thiazolidinediones within 3 months, or any other drugs for treatment of hyperglycemia (except metformin) within 2 months, prior to the first week of the study
* Have hepatitis B and/or positive hepatitis B surface antigen. hepatitis C or human immunodeficiency virus (HIV) and/or positive HIV antibodies
* Have known or suspected cardiac autonomic neuropathy (for example, resting tachycardia or orthostatic hypotension), based on clinical signs, symptoms, or appropriate diagnostic testing
* Have cardiac disease with functional status that is New York Heart Association Class II, III, or IV or in the last 6 months have had any of the following: a history of myocardial infarction , unstable angina, coronary artery bypass graft, percutaneous coronary intervention (diagnostic angiograms are permitted), transient ischemic attack, or cerebrovascular accident (for example, stroke)
* Have poorly controlled hypertension, malignant hypertension, renal artery stenosis, and/or evidence of labile blood pressure including symptomatic postural hypotension. Doses of antihypertensive medications must be stable for 30 days prior to the first week of the study
* Have obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis, or an alanine transaminase or aspartate aminotransferase levels >2 times the upper limit of the reference range
* Have evidence of hypothyroidism or hyperthyroidism based on clinical evaluation and/or an abnormal thyroid-stimulating hormone which, in the opinion of the investigator, would pose a risk to participant safety. Participants on a stable dose of thyroid replacement therapy may be eligible if they meet the other criteria
* Have clinically significant peripheral vascular disease, or clinical evidence of active diabetic proliferative retinopathy, (known significant autonomic neuropathy) as evidenced by urinary retention, orthostatic hypotension, diabetic diarrhea or gastroparesis
* Have an active or untreated malignancy or have been in remission from a clinically significant malignancy (other than basal or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for less than 5 years
* Have impaired renal function
* Have fasting triglycerides >500 milligrams per deciliter (mg/dL) at screening
* Have experienced a keto-acidotic episode requiring hospitalization in the last 6 months
* Have an electrocardiogram (ECG) considered to be indicative of cardiac disease
* Have personal or family history of long QT syndrome, family history of sudden death in a first-degree relative before age 40, or personal history of unexplained syncope within the last year. Use of prescription or over-the-counter medications known to prolong the QT or QTc interval
* Have a history of bone disease (including osteoporosis or unhealed fractures), evidence of osteoporosis (femoral neck or lumbar spine T-score <-2.5) determined by dual X-ray absorptometry (DXA) scan at screening, evidence of osteopenia (T-score between -1.0 and -2.5 at the femoral neck or lumbar spine) with a high risk of fracture based on risk factors or current active treatment of periodontal disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM -5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - Orange County Research Center, Orange, California
  - Miami Research Associates, Miami, Florida
  - Compass Research, Orlando, Florida
  - Clinilabs, Inc (New York), New York, New York
  - Dallas Diabetes Endocrine Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was planned in 2 stages; Stage 1 evaluated up to 5 escalating parallel-dose groups. Stage 2, which was to evaluate participants stratified by Hemoglobin A1c (HbA1c), metformin therapy, and washout of a second oral anti-hyperglycemic medication (OAM) was not conducted because of inadequate efficacy at well-tolerated doses in Stage 1.
Groups:
- Placebo: Placebo administered by subcutaneous injection (SC) once a week (Q1W) for 12 weeks
- 7 mg LY3053102: 7 mg LY3053102 administered SC Q1W for 12 weeks.
- 15 mg LY3053102: 15 mg LY3053102 administered SC Q1W for 12 weeks.
- 50 mg LY3053102: 50 mg LY3053102 administered SC Q1W for 12 weeks.
- 100 mg LY3053102: 100 mg LY3053102 administered SC Q1W for 12 weeks.
- 200 mg LY3053102: 200 mg LY3053102 administered SC Q1W for 12 weeks.
- 2 mg Exenatide ER: 2 mg exenatide ER administered SC Q1W for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | 7 mg LY3053102 | 15 mg LY3053102 | 50 mg LY3053102 | 100 mg LY3053102 | 200 mg LY3053102 | 2 mg Exenatide ER
Started | 10 | 8 | 8 | 8 | 8 | 8 | 10
Received at Least One Dose of Study Drug | 10 | 8 | 8 | 7 | 8 | 8 | 10
Completed | 10 | 7 | 6 | 6 | 6 | 3 | 6
Not Completed | 0 | 1 | 2 | 2 | 2 | 5 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 1 | 1 | 0
Not completed — Early Termination Criteria Met | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Randomized in Error | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Placebo: Placebo administered SC QW for 12 weeks
- 7 mg LY3053102: 7 mg LY3053102 administered SC QW for 12 weeks
- 15 mg LY3053102: 15 mg LY3053102 administered SC QW for 12 weeks
- 50 mg LY3053102: 50 mg LY3053102 administered SC QW for 12 weeks
- 100 mg LY3053102: 100 mg LY3053102 administered SC QW for 12 weeks
- 200 mg LY3053102: 200 mg LY3053102 administered SC QW for 12 weeks
- 2 mg Exenatide ER: 2 mg Exenatide ER administered SC QW for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | 7 mg LY3053102 | 15 mg LY3053102 | 50 mg LY3053102 | 100 mg LY3053102 | 200 mg LY3053102 | 2 mg Exenatide ER | Total
Number analyzed (Participants) | 10 | 8 | 8 | 7 | 8 | 8 | 10 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.9 (8.9) | 57.3 (4.9) | 59.9 (5.8) | 56.3 (6.0) | 50.8 (13.0) | 54.6 (8.3) | 52.8 (9.1) | 55.3 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 4 | 2 | 4 | 4 | 2 | 24
  Male | 5 | 5 | 4 | 5 | 4 | 4 | 8 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 3 | 5 | 6 | 8 | 2 | 35
  Not Hispanic or Latino | 3 | 4 | 5 | 2 | 2 | 0 | 8 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 4 | 2 | 2 | 0 | 3 | 11
  White | 10 | 7 | 4 | 5 | 6 | 8 | 4 | 44
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 8 | 8 | 7 | 8 | 8 | 10 | 59
Baseline Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent of HbA1c] | 8.39 (0.80) | 8.33 (1.17) | 7.93 (0.81) | 8.30 (0.74) | 9.40 (1.43) | 8.10 (0.63) | 8.50 (1.03) | 8.42 (1.02)
Baseline Fasting Plasma Glucose [Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)] | 180.6 (45.3) | 178.6 (44.3) | 176.6 (58.0) | 173.3 (39.6) | 183.3 (46.2) | 185.9 (50.6) | 150.6 (46.8) | 174.9 (46.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at 12-Week Endpoint
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) analysis adjusting for metformin use, washout of second oral anti-hyperglycemic medication (OAM), treatment, visit, and treatment-by-visit interaction as fixed effects, baseline as a covariate, and participant as a random effect.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug, and who had baseline and post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: Percent of HbA1c
Groups:
- Placebo: Placebo administered SC Q1W for 12 weeks
Arm/Group | Placebo | 7 mg LY3053102 | 15 mg LY3053102 | 50 mg LY3053102 | 100 mg LY3053102 | 200 mg LY3053102 | 2 mg Exenatide ER
Number analyzed (Participants) | 10 | 7 | 5 | 5 | 7 | 3 | 6
Percent of HbA1c | -0.49 (0.33) | -0.70 (0.40) | -0.75 (0.44) | -0.22 (0.43) | -0.48 (0.40) | -0.52 (0.47) | -1.43 (0.36)

2. Secondary Outcome: Percentage of Participants Achieving HbA1c <7.0% or HbA1c ≤6.5% at 12-Week Endpoint
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time.
Time Frame: Week 12
Population: All randomized participants who received at least 1 dose of study drug, and who had baseline and post-baseline data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 7 mg LY3053102 | 15 mg LY3053102 | 50 mg LY3053102 | 100 mg LY3053102 | 200 mg LY3053102 | 2 mg Exenatide ER
Number analyzed (Participants) | 10 | 8 | 8 | 7 | 8 | 8 | 10
Percentage of Participants
  HbA1c <7.0%: number analyzed (Participants) | 10 | 7 | 5 | 5 | 7 | 3 | 6
  HbA1c <7.0% | 0.0 | 14.3 | 40.0 | 20.0 | 0.0 | 0.0 | 83.3
  HbA1c ≤6.5%: number analyzed (Participants) | 10 | 7 | 5 | 5 | 7 | 3 | 6
  HbA1c ≤6.5% | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 66.7

3. Secondary Outcome: Percentage of Participants That Require Rescue Therapy
Description: Percentage of participants that required >=1 rescue (blood glucose lowering) medications.
Time Frame: Baseline through Week 12
Population: All randomized participants who took at least 1 dose of study drug, and who had a baseline and a post-baseline measurement for the time point.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 7 mg LY3053102 | 15 mg LY3053102 | 50 mg LY3053102 | 100 mg LY3053102 | 200 mg LY3053102 | 2 mg Exenatide ER
Number analyzed (Participants) | 10 | 8 | 8 | 7 | 8 | 8 | 10
Percentage of Participants | 0.0 | 0.0 | 12.5 | 14.3 | 0.0 | 0.0 | 0.0

4. Secondary Outcome: Change From Baseline in Body Weight at 12-Week Endpoint
Description: LS means were calculated using MMRM analysis adjusting for baseline HbA1c category, metformin use, washout of second OAM, treatment, visit, and treatment-by-visit interaction as fixed effects, baseline as a covariate, and participant as a random effect (excludes data after rescue therapy).
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug, and who had baseline and post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Groups:
- 50 mg LY3053102: 50 mg LY3053102 50 mg administered SC Q1W for 12 weeks
Arm/Group | Placebo | 7 mg LY3053102 | 15 mg LY3053102 | 50 mg LY3053102 | 100 mg LY3053102 | 200 mg LY3053102 | 2 mg Exenatide ER
Number analyzed (Participants) | 10 | 7 | 5 | 5 | 7 | 4 | 7
kilogram (kg) | 0.7 (1.1) | 1.5 (1.3) | 0.0 (1.4) | 0.4 (1.4) | -1.7 (1.3) | -2.0 (1.4) | -0.1 (1.1)

5. Secondary Outcome: Change From Baseline in 7-Point Blood Glucose Profile at 12-Week Endpoint
Description: 7-Point Self-Monitored Blood Glucose profiles are measures of blood glucose concentration taken 7 times a day at morning pre-prandial, morning 2 hours postprandial, midday pre-prandial, midday 2 hours postprandial, evening pre-prandial, evening 2 hour postprandial, and bedtime. LS means were calculated using MMRM analysis adjusting for baseline HbA1c category, metformin use, washout of second OAM, treatment, visit, and treatment-by-visit interaction as fixed effects, baseline as a covariate, and participant as a random effect (excludes data after rescue therapy).
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug, and who had baseline and post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: milligram/deciliter (mg/dL)
Arm/Group | Placebo | 7 mg LY3053102 | 15 mg LY3053102 | 50 mg LY3053102 | 100 mg LY3053102 | 200 mg LY3053102 | 2 mg Exenatide ER
Number analyzed (Participants) | 10 | 7 | 5 | 5 | 7 | 3 | 5
milligram/deciliter (mg/dL)
  Morning Meal (Post- minus Pre-prandial) | -23.4 (15.8) | -18.7 (19.4) | -57.7 (21.6) | -34.9 (21.9) | 4.7 (18.3) | -26.8 (25.8) | -47.9 (19.4)
  Midday Meal (Post- minus Pre-prandial) | -1.1 (22.4) | -31.3 (27.5) | -55.0 (29.2) | -24.7 (29.2) | 2.5 (25.8) | -24.6 (32.3) | -31.3 (24.9)
  Evening Meal (Post- minus Pre-prandial) | -18.8 (20.8) | -11.1 (25.8) | -46.5 (27.5) | -25.9 (27.9) | -39.0 (24.1) | -61.3 (31.4) | -4.9 (24.2)
  Bedtime | 3.9 (19.1) | 18.8 (23.3) | -44.5 (28.1) | -10.1 (25.7) | 4.9 (22.1) | -13.0 (30.8) | -53.6 (23.5)

6. Secondary Outcome: Change From Baseline in Lipids at 12-Week Endpoint
Description: Lipids includes: High Density Lipoprotein-Cholesterol (HDL-C), Low Density Lipoprotein-Cholesterol (LDL-C), Triglycerides, and Cholesterol. LS means were calculated using MMRM analysis adjusting for metformin use, washout of second OAM, baseline HbA1c category, treatment, visit, and treatment-by-visit interaction as fixed effects, baseline as a covariate, and participant as a random effect (excludes data after rescue therapy).
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug, and who had baseline and post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | 7 mg LY3053102 | 15 mg LY3053102 | 50 mg LY3053102 | 100 mg LY3053102 | 200 mg LY3053102 | 2 mg Exenatide ER
Number analyzed (Participants) | 10 | 8 | 8 | 7 | 8 | 8 | 10
mg/dL
  HDL-C: number analyzed (Participants) | 10 | 7 | 5 | 5 | 7 | 4 | 7
  HDL-C | 1.0 (2.2) | 6.0 (2.6) | 9.3 (2.9) | 6.4 (2.9) | 6.0 (2.6) | 11.4 (3.1) | -2.3 (2.2)
  LDL-C: number analyzed (Participants) | 9 | 7 | 5 | 5 | 7 | 4 | 7
  LDL-C | 12.1 (10.4) | 6.8 (12.0) | -25.6 (13.8) | -6.5 (13.5) | -2.2 (12.0) | -7.3 (14.5) | -19.9 (11.3)

7. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies to LY3053102
Description: Percentage of participants with anti-LY3053102 antibody titre changes from baseline to the maximum postbaseline value.
Time Frame: Baseline through Study Completion (Up to 6 Months)
Population: All randomized participants who received at least 1 dose of study drug and had evaluable immunogenicity.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 7 mg LY3053102 | 15 mg LY3053102 | 50 mg LY3053102 | 100 mg LY3053102 | 200 mg LY3053102 | 2 mg Exenatide ER
Number analyzed (Participants) | 10 | 8 | 8 | 7 | 8 | 8 | 10
Percentage of Participants | 0 | 1 | 1 | 0 | 2 | 2 | 2

8. Secondary Outcome: Percentage of Participants With Hypoglycemia
Description: Hypoglycemia was defined as any event meeting the criteria for documented symptomatic hypoglycemia, asymptomatic hypoglycemia, or probable symptomatic hypoglycemia.
Time Frame: Baseline through Week 12
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 7 mg LY3053102 | 15 mg LY3053102 | 50 mg LY3053102 | 100 mg LY3053102 | 200 mg LY3053102 | 2 mg Exenatide ER
Number analyzed (Participants) | 10 | 8 | 8 | 7 | 8 | 8 | 10
Percentage of Participants | 10.0 | 12.5 | 0.0 | 0.0 | 12.5 | 12.5 | 20.0

9. Secondary Outcome: Change From Baseline in Bone Metabolism at 12-Week Endpoint (Osteocalcin and Bone-Specific Alkaline Phosphatase [Bone-Specific ALP])
Description: LS means were calculated using MMRM analysis adjusting for metformin use, washout of second OAM, baseline HbA1c category, treatment, visit, and treatment-by-visit interaction as fixed effects, baseline as a covariate, and participant as a random effect (excludes data after rescue therapy).
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: microgram/liter (ug/L)
Arm/Group | Placebo | 7 mg LY3053102 | 15 mg LY3053102 | 50 mg LY3053102 | 100 mg LY3053102 | 200 mg LY3053102 | 2 mg Exenatide ER
Number analyzed (Participants) | 10 | 8 | 8 | 7 | 8 | 8 | 10
microgram/liter (ug/L)
  Osteocalcin: number analyzed (Participants) | 10 | 7 | 6 | 6 | 7 | 4 | 7
  Osteocalcin | 1.2 (1.1) | -0.7 (1.3) | -1.7 (1.3) | 0.0 (1.4) | -2.6 (1.2) | -0.2 (1.4) | 0.3 (1.0)
  Bone-Specific ALP: number analyzed (Participants) | 10 | 7 | 6 | 6 | 7 | 4 | 7
  Bone-Specific ALP | 0.4 (0.8) | -0.1 (0.9) | -0.2 (1.0) | -1.9 (1.0) | -1.9 (0.9) | -0.3 (1.0) | -2.3 (0.7)

10. Secondary Outcome: Change From Baseline in Bone Metabolism at 12-Week Endpoint (Beta-Crosslaps and Procollagen 1 N-Terminal Propeptide [P1NP])
Description: as for outcome 9
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: nanogram/milliliter (ng/mL)
Arm/Group | Placebo | 7 mg LY3053102 | 15 mg LY3053102 | 50 mg LY3053102 | 100 mg LY3053102 | 200 mg LY3053102 | 2 mg Exenatide ER
Number analyzed (Participants) | 10 | 8 | 8 | 7 | 8 | 8 | 10
nanogram/milliliter (ng/mL)
  Beta-Crosslaps: number analyzed (Participants) | 10 | 7 | 6 | 6 | 7 | 4 | 7
  Beta-Crosslaps | -0.038 (0.042) | -0.033 (0.052) | -0.023 (0.051) | 0.001 (0.053) | 0.004 (0.048) | 0.031 (0.054) | -0.010 (0.040)
  P1NP: number analyzed (Participants) | 10 | 7 | 6 | 6 | 7 | 4 | 6
  P1NP | 5.0 (2.8) | -0.3 (3.4) | 0.9 (3.5) | 1.9 (3.5) | -6.8 (3.2) | -0.2 (3.8) | 2.3 (2.9)

11. Secondary Outcome: Change From Baseline in Bone Mineral Density Markers at 12-Week Endpoint
Description: as for outcome 9
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: milligram/square centimeter (mg/cm2)
Arm/Group | Placebo | 7 mg LY3053102 | 15 mg LY3053102 | 50 mg LY3053102 | 100 mg LY3053102 | 200 mg LY3053102 | 2 mg Exenatide ER
Number analyzed (Participants) | 10 | 8 | 8 | 7 | 8 | 8 | 10
milligram/square centimeter (mg/cm2)
  L1-L4 Intervertebral Space: number analyzed (Participants) | 10 | 7 | 7 | 6 | 8 | 5 | 9
  L1-L4 Intervertebral Space | 1.4 (1.6) | -0.4 (1.9) | 1.2 (2.0) | 1.0 (2.1) | 2.0 (1.8) | 1.6 (2.1) | 1.8 (1.4)
  Neck of Femur: number analyzed (Participants) | 10 | 7 | 6 | 6 | 8 | 5 | 9
  Neck of Femur | 0.2 (1.6) | -0.6 (1.9) | -0.4 (2.0) | -0.8 (2.0) | -0.3 (1.8) | -1.2 (2.1) | -2.1 (1.4)
  Total Hip: number analyzed (Participants) | 10 | 7 | 6 | 6 | 8 | 5 | 9
  Total Hip | 0.2 (1.0) | -0.6 (1.2) | -0.7 (1.2) | -1.0 (1.2) | 0.1 (1.1) | -0.7 (1.3) | -1.0 (0.8)

12. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve During One Dosing Interval at Steady State (AUC [τ,ss]) of LY3053102
Description: AUC (τ,ss) = area under the concentration versus time curve during one dosing interval at steady state, where the dosing interval (τ) = 168 hours.
Time Frame: Predose, 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 168 hours post-dose
Population: All randomized participants who received at least 1 dose of study drug and had evaluable pharmacokinetics
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram•hour/milliliter (µg•h/mL)
Arm/Group | 7 mg LY3053102 | 15 mg LY3053102 | 50 mg LY3053102 | 100 mg LY3053102 | 200 mg LY3053102
Number analyzed (Participants) | 8 | 8 | 7 | 8 | 8
microgram•hour/milliliter (µg•h/mL) | 22.6 (32.1) | 76.8 (25.6) | 190.0 (47.3) | 350.0 (36.3) | 917.0 (35.1)

ADVERSE EVENTS:
Description: One participant was discontinued from the study before dosing due to meeting exclusion criteria.
Groups:
- Placebo: Placebo administered by SC QW for 12 weeks
Arm/Group | Placebo | 7 mg LY3053102 | 15 mg LY3053102 | 50 mg LY3053102 | 100 mg LY3053102 | 200 mg LY3053102 | 2 mg Exenatide ER
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/8 | 0/8 | 0/7 | 1/8 | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 4/8 | 4/8 | 4/7 | 7/8 | 7/8 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | 7 mg LY3053102 (N=8) | 15 mg LY3053102 (N=8) | 50 mg LY3053102 (N=7) | 100 mg LY3053102 (N=8) | 200 mg LY3053102 (N=8) | 2 mg Exenatide ER (N=10)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | 7 mg LY3053102 (N=8) | 15 mg LY3053102 (N=8) | 50 mg LY3053102 (N=7) | 100 mg LY3053102 (N=8) | 200 mg LY3053102 (N=8) | 2 mg Exenatide ER (N=10)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 6 (9) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (6) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 4 (5) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site discolouration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site erosion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 1 (3) | 4 (7) | 1 (1)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site nodule (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (4) | 2 (2) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site urticaria (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 5 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac stress test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (8)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 3 (3) | 4 (5) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypogeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Stage 2, which was to evaluate participants stratified by HbA1c, metformin therapy, and washout of a second oral anti-hyperglycemic medication (OAM) was not conducted because of inadequate efficacy at well-tolerated doses in Stage 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days